CLINICAL TRIAL: NCT02983760
Title: Comparison of 3 Diagnostic Strategies of Pulmonary Embolism : Planar Ventilation-perfusion Scintigraphy (Planar V/Q Scan), Computed Tomography Pulmonary Angiography (CTPA), and V/Q Single Photon Emission Computed Tomography (SPECT)
Brief Title: Comparison of 3 Diagnostic Strategies of PE: Planar V/Q Scan, CTPA, and V/Q SPECT.
Acronym: SPECTACULAR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The enrollment process for patients is difficult.
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SPECTACULAR - RB 16.068
Record Dates: First submitted 2016-11-28; First posted 2016-12-06 (Estimated); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Pulmonary Embolism
Keywords: Pulmonary embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Planar V/Q-based strategy (Active Comparator): Control arm
  Interventions: Device: Planar V/Q-based strategy
- CTPA-based strategy (Active Comparator): Control arm
  Interventions: Device: CTPA-based strategy
- V/Q SPECT-based strategy (Experimental): Experimental arm
  Interventions: Device: V/Q SPECT-based strategy

INTERVENTIONS:
Device: Planar V/Q-based strategy — Strategy based on planar pulmonary scintigraphy
  Arms: Planar V/Q-based strategy
Device: CTPA-based strategy — Strategy based on pulmonary angiography
  Arms: CTPA-based strategy
Device: V/Q SPECT-based strategy — Strategy based on pulmonary tomoscintigraphy
  Arms: V/Q SPECT-based strategy

SUMMARY:
Pulmonary embolism (PE) remains a diagnostic challenge. False negative testing exposes patient to the risk of potentially fatal recurrence. False positive testing exposes patients to potentially fatal unduly side effects of anticoagulants.

Current diagnostic strategies rely on the sequential use of pretest clinical probability, Ddimer test, and chest imaging. Two chest imaging modalities have been validated for PE diagnostic exclusion: Computed Tomography Pulmonary Angiography (CTPA) and planar V/Q scan. Main limitations of planar V/Q are the high proportion of non-conclusive results, therefore requiring additional testing and more complex diagnostic algorithms. Main limitations of CTPA are its higher radiation dose and contraindications (renal failure).

In a randomized trial that compared strategies based on CTPA and on planar V/Q scan, a 30% increase in the rate of PE diagnoses was found in the arm using CTPA, raising the hypothesis of over-diagnosing and over-treating PE when using CTPA.

V/Q Single Photon Emission CT (SPECT) is a new method of scintigraphic acquisition that has been reported to improve the diagnostic performances of the test, which could reduce the number of non-conclusive tests and allow simplified diagnostic algorithms.

The investigators hypothesize that a strategy based on V/Q SPECT could be an alternative to the two usual approaches responding rightly to the two mains issues and combining the advantages of CTPA (simplified diagnostic approach) and planar V/Q (no overdiagnosis, lower radiation exposure, no contraindication).

Although a recent survey showed that up to 70% of nuclear medicine centers perform SPECT rather than planar imaging for diagnosing PE, a diagnostic management outcome study, in which diagnostic decision would be made on the basis of a standardized algorithm based on the V/Q SPECT is lacking. Such a study needs to be conducted to ensure that the safety of diagnostic exclusion using a V/Q SPECT based strategy is non-inferior to that of previously validated strategies, and to verify that the use of V/Q SPECT does not lead to over-diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with a clinically suspected PE (defined as an acute onset of new or worsening shortness of breath, chest pain, hemoptysis, presyncope, or syncope) without another obvious apparent cause.
* High pretest clinical probability of PE or a non-high pretest clinical probability but a positive D-Dimer test.

Exclusion Criteria:

* Age less than 18 years
* Patients with already confirmed PE
* Patients with a clinically suspected high-risk pulmonary embolism (hypotension or shock)
* Use of therapeutic doses of anticoagulants for more than 48 hours
* Other indication for long-term use of anticoagulants
* Contraindication to contrast media (including renal insufficiency with a creatinine clearance lower than 30 ml/min)
* Life expectancy less than 3 months
* Unable/unwilling to give informed consent
* Unlikely to comply with study follow-up
* Ongoing pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 611 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2024-12-17 (Actual); Study Completion 2024-12-17 (Actual)

PRIMARY OUTCOMES:
Thromboembolic events rate in a 3 month follow-up period in patients left untreated after a negative diagnostic strategy. | 3 months
  Rate of symptomatic objectively confirmed thromboembolic events during the 3-month follow-up period in patients left untreated after a negative diagnostic work-up in V/Q SPECT-based strategy in comparison with planar V/Q-based strategy and CTPA-based strategy.

SECONDARY OUTCOMES:
Proportion of PE diagnostic in each arm | 3 months
  Proportion of patients deemed to have PE according to the strategy in each arm.
Proportion of additionnal tests required in each arm | 3 months
  Proportion of patients for whom additional tests are requested in each arm.
Major bleeding incidence in each arm | 3 months
  Incidence of major bleeding episodes in each arm.
Incidence and cause of death in each arm | 3 months
  Incidence and cause of death in each arm

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Yves Salaun, Study Director — CHRU de Brest
Locations (11):
- Ottawa, Ottawa, Canada
- France (9):
  - Hopital Saint Esprit, Agen
  - CHU d'ANGERS, Angers
  - CHRU de Brest, Brest
  - CHU Clermont Ferrand, Clermont-Ferrand
  - CH des Pays de Morlaix, Morlaix
  - Hegp - Ap-Hp, Paris
  - CHU la Réunion, Saint-Denis
  - CHU de Saint Etienne, Saint-Etienne
  - CH Toulon, Toulon
- Geneva University Hospital, Geneva, Switzerland

REFERENCES:
- [Derived] Le Pennec R, Le Roux PY, Robin P, Couturaud F, Righini M, Le Gal G, Salaun PY. Comparison of three diagnostic strategies for suspicion of pulmonary embolism: planar ventilation-perfusion scan (V/Q), CT pulmonary angiography (CTPA) and single photon emission CT ventilation-perfusion scan (SPECT V/Q): a protocol of a randomised controlled trial. BMJ Open. 2024 May 15;14(5):e075712. doi: 10.1136/bmjopen-2023-075712. PMID 38754880